CLINICAL TRIAL: NCT05346315
Title: Registered Dietitian Nutritionist Led Food as Medicine Program in the Food Retail Setting: A Feasibility Study
Brief Title: Food as Medicine Study
Acronym: FaM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Other Study IDs: 1329215
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Nutrition Disorders
Keywords: Dietitian; Feasibility; E-commerce
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RDN Medical Nutrition Therapy — The RDNs will provide bi-monthly nutrition care, counseling, and dietary recommendations for a 6-month intervention, delivered either in-person or via telehealth, to the grocery store patrons during the study intervention. The RDN will provided care to the participant based upon the participant's unique dietary and nutritional needs. The RDN will provide nutrition recommendations and create meal plans via NutriStyle for the participants to follow. The meal plans will be uploaded into the grocery store's E-commerce shopping platform, which the participant can utilize to purchase foods that are needed to follow the RDNs nutrition recommendations for an individual person.

SUMMARY:
The purpose of this study is to demonstrate proof of concept that registered dietitian nutritionists (RDNs) can implement a Food as Medicine program that utilizes a grocery E-commerce platform in a food retail setting, and the process of measuring the outcomes is feasible.

DETAILED DESCRIPTION:
The Academy of Nutrition and Dietetics Data Science Center (DSC) will implement the proposed prospective feasibility study. The study aims to measure change in nutrition problems, eating patterns, food purchasing patterns and health outcomes of participants who have agreed to receive a 6-month RDN-led Food as Medicine intervention program in the food retail setting. The intervention will be provided to all study participants and change will be evaluated in participants by comparing data at baseline and endline. The Food as Medicine intervention program will consist of:

* Personalized nutrition counseling (delivered in-person or telehealth, depending on preferences of the participant) by Hy-Vee RDNs.
* Personalized meal plans (based on program participants' individual anthropometrics, disease state, health goals, culture, food allergies / intolerances and eating preferences). The meal plans will be generated by the nutrition technology software, NutriStyle.
* Personalized shopping lists generated by a nutrition technology software (NutriStyle) and utilized for in-store grocery shopping, online grocery pick-up or online grocery delivery.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old
2. Household/participant willing to utilize the shopping list provided
3. No new medical diagnoses or medications (unrelated to the study intervention) within the last 3 months and no anticipated changes during the intervention period. (The participant may have a new medical diagnosis for which they are seeking MNT.)
4. Nebraska or Iowa resident
5. Minimum of one new self-reported diagnosis or an existing diagnosis that participant has not sought MNT for previously: Overweight/obesity, Hypertension, Cardiovascular disease, Pre-diabetes, Type 2 diabetes
6. First visit with the RDN for the current medical diagnosis (may have received MNT for other conditions previously)
7. Access to Hy-Vee Aisles Online and NutriStyle, through the computer or mobile app
8. Willing to use Hy-Vee's Aisles Online e-commerce platform and NutriStyle
9. Willing to meet with a Hy-Vee RDN regularly in person or via telehealth (and talk on the phone with the Hy-Vee RDN monthly) throughout the study intervention (6 months)
10. Current Hy-Vee fuel saver card holder, or willing to obtain a fuel saver card
11. Provide verbal and written communication and written informed consent in English

Exclusion Criteria:

1. Prescribed or taking over-the-counter weight loss medication at enrollment
2. Prescribed corticosteroids or other drug known to interfere with glucose metabolism
3. Scheduled for bariatric weight loss surgery during 6-month study intervention period
4. Pregnant/lactating
5. Currently working with another nutrition care professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 18 years old; a resident of Nebraska or Iowa; have at least 1 of the following diagnoses that the person is not received nutrition counseling for: overweight / obesity, hypertension, cardiovascular disease, type 2 diabetes, or pre-diabetes; and willing to follow a meal plan and order groceries through Hy-Vee Aisles Online for 6-months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in resolution of nutrition problem | 6 months
  Percent of resolution of nutrition problems
Change in eating pattern score | 6 months
  Picture your Plate Survey (Score ranges from minimum 0 to maximum 96 with 96 being the best score)

SECONDARY OUTCOMES:
Change in body weight | 6 months
  pounds
Change in Body Mass Index (BMI) | 6 months
  kg/m2
Change in waist circumference | 6 months
  inches
Change in total cholesterol (LDL, HDL, Triglycerides) | 6 months
  mg/dL
Change in fasting blood glucose | 6 months
  mg/dL
Change in blood pressure (systolic and diastolic) | 6 months
  mmHg
Change in basket size | 6 months
  Dollars spent per order
Change in perceived shopping list adherence | 6 months
  Perceived compliance score (Score ranges from 1 minimum to 10 maximum with 10 being the best score)
Change in shopping frequency | 6 months
  # orders place in the 6 month period vs. previous 6 months
Change in health quality of life | 6 months
  CDC's Health Related Quality of Life-14 Survey (Score is determined by overall healthy days vs. unhealthy days in a given month)

CONTACTS AND LOCATIONS:
Overall Officials: Constantina Papoutsakis, PhD, RD, Principal Investigator — Academy of Nutrition and Dietetics
Locations (3):
- United States (3):
  - Amber Pharmacy, Omaha, Nebraska
  - Linden Market Hy-Vee, Omaha, Nebraska
  - Papillion Hy-Vee, Papillion, Nebraska

IPD SHARING:
Plan to Share IPD: No